CLINICAL TRIAL: NCT05074173
Title: Simple Text-Messaging and Social Support to Increase Hypertension Medication Adherence in New Orleans, Louisiana (LA)
Brief Title: Text My Hypertension BP Meds NOLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: LA CaTS Clinical Research Resources Core (Unknown); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-887; 5U54GM104940-05 (NIH)
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Hypertension
Keywords: Quality of life; Adherence; High blood pressure
MeSH Terms: conditions — Hypertension | interventions — Communication Devices for People with Disabilities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Group (Other): Participants will be enrolled in a bidirectional text messaging system from Tulane University Medical Group where they will receive and send text from their mobile phones to monitor their anti-hypertension medication regimen. Text messages will be sent: daily for medication and refill reminders; weekly for hypertension education messages and asking if a support person helped them with medication reminders. Study personnel will educate participants on proper blood pressure technique to conduct self-measured blood pressure (SMBP) at home. These blood pressure values will be automatically uploaded twice daily from a Bluetooth device to a phone application to allow the participant and healthcare team track their blood pressure. Participants will receive the Bluetooth blood pressure device to perform SMBP at enrollment.
  Interventions: Behavioral: Text

INTERVENTIONS:
Behavioral: Text — These blood pressure values will be automatically uploaded twice daily from a Bluetooth device to a phone application to allow the participant and healthcare team track their blood pressure.

SUMMARY:
The specific aims of this research study are to

1. Engage participants with poorly controlled hypertension and medication non-adherence to use simple digital approaches, specifically recurring text-messages to improve medication adherence.
2. Promote participant medication adherence and interaction with telehealth platforms with recurring text reminders on medication schedules and refills, science-based hypertension education content, and communication exchange with their health providers to improve blood pressure.
3. Evaluate the role of social support in helping participants manage their hypertension and control of Cardiovascular disease (CVD) risk factors, including daily blood pressure measurement, changes in participant quality of life, and barriers towards medication adherence, and setting goals for health behaviors.

DETAILED DESCRIPTION:
All eligible participants will be enrolled into the study at the Tulane cardiology clinic for an 8-week period. Key study personnel will screen patients from the clinic interested in the study during their appointment visit. Identifying information that will be collected from participants will be name, date of birth, and telephone number to send them text messages. Potential participants making study inquiries by email will receive prompt responses. If the participant does not enroll in the study because they are not eligible, the information will be shredded. Study personnel will also review medical records of Dr. Keith Ferdinand to identify potential patients and provide the subjects with study information (e.g. flyers, advertisements, recruitment script, etc.) The subjects may then approach the study team about participation. Study personnel will arrange a time and date with the church community site to distribute flyers describing the study to church congregants to seek study interest. Interested persons can be screened on-site for eligibility or at a date to be determined by congregants. Study personnel will use an eligibility checklist to screen participants.

Below are procedures performed during the study and the time expected to complete each task:

This study will follow an 8-week interventional cohort design using a series of questionnaires to collect data pre-post study procedures from two sites: Tulane cardiology clinic and Christian Unity Baptist Church. Participants will be screened for eligibility at both sites by in-person interviews, telephone using an Institutional Review Board (IRB) approved recruitment script, and/or clinic medical records. After screening, eligible participants will be enrolled into the study at Tulane cardiology clinic by study personnel. Blood pressure and weight will be measured by study personnel on the first and the last day of the study, in addition to calculating their risk for heart attack and stroke using the Atherosclerotic cardiovascular disease (ASCVD) Risk Estimator Plus.

9 Study personnel will calculate participant's ASCVD risk by downloading the app on their mobile device. No patient information is collected and stored in the app. Anonymous user behavior (e.g., number of people who downloaded the app, how many times a day the app was used) will be gathered through Google Analytics. All data collected in the app is anonymous and cannot be traced back to an individual user.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years of age.
* Speak and read English.
* Diagnosis of stage 1* and 2** hypertension (HTN), taking at least one antihypertensive medication.
* Internet and mobile phone access with two-way texting capability.
* > 1 on 4-item Krousel-Wood Medication Adherence Scale (K-Wood-MAS-4) or similar tool.
* Able to download blood pressure tracking App to mobile phone. (*Stage 1 HTN: 130-139 mmHg or 80-89 mmHg16) (**Stage 2 HTN: 140 mmHg or higher or >90 mmHg16)

Exclusion Criteria:

* Having been hospitalized within 6 months of starting the study if the patient has a diagnosis of heart failure, end-stage kidney disease, acute coronary syndrome, or stroke.
* Plans to cancel mobile phone plan within 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-05-28 (Actual); Study Completion 2022-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Ferdinand, MD, Principal Investigator — Tulane University School of Medicine
Locations (2):
- United States (2):
  - Christian Unity Baptist Church, New Orleans, Louisiana
  - Tulane University Medical Center, New Orleans, Louisiana

REFERENCES:
- [Background] Ferdinand KC, Senatore FF, Clayton-Jeter H, Cryer DR, Lewin JC, Nasser SA, Fiuzat M, Califf RM. Improving Medication Adherence in Cardiometabolic Disease: Practical and Regulatory Implications. J Am Coll Cardiol. 2017 Jan 31;69(4):437-451. doi: 10.1016/j.jacc.2016.11.034. PMID 28126162
- [Background] Ferdinand DP, Nedunchezhian S, Ferdinand KC. Hypertension in African Americans: Advances in community outreach and public health approaches. Prog Cardiovasc Dis. 2020 Jan-Feb;63(1):40-45. doi: 10.1016/j.pcad.2019.12.005. Epub 2019 Dec 19. PMID 31863786

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patient Group
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patient Group
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.68 (12.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 32
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 36
Type 2 Diabetes [Count of Participants; unit: Participants]
  Yes | 26
  No | 9
  Unknown | 1
Obesity [Count of Participants; unit: Participants]
  Obese | 26
  Not Obese | 10

OUTCOME MEASURES:

1. Primary Outcome: Measure of Quality of Life Assessed by 14-item Center for Disease Control (CDC) Health Related Quality of Life Questioner
Description: The change of quality of life will be measured by the responses from the 14-item Center for Disease Control (CDC) Health Related Quality of Life questioner at the enrollment (baseline) visit and at the end of study visit at 2 months. The questioner is a CDC designed quality of life survey that has 14 questions, and the investigators calculated the unhealthy days score for each participant.
  Unhealthy days are an estimate of the overall number of days during the previous 30 days when the respondent felt that either his or her physical or mental health was not good. To obtain that estimate, responses to questions 2 and 3 were combined to calculate a summary index of overall unhealthy days with a logical maximum of 30 unhealthy days. The range is from 0 to 30, minimum would be 0 which indicates better outcome and 30 is the maximum and would indicate poor outcome.
Time Frame: Baseline, 2 months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Patient Group
Number analyzed (Participants) | 36
Days
  Baseline | 9.11 (10.36)
  2 Months | 6.81 (9.89)

2. Secondary Outcome: Change in Systolic and Diastolic Blood Pressure Done by Investigators
Description: Change in systolic and diastolic blood pressure, which was done using 2 seated blood pressure readings using validated approaches, measured in millimeters of mercury from day one of enrollment (baseline) and at end of study visit.
Time Frame: Baseline, 2 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Patient Group
Number analyzed (Participants) | 36
mmHg
  Systolic blood pressure at baseline | 142.19 (18.94)
  Systolic blood pressure at 2 months | 131.69 (13.99)
  Diastolic blood pressure at baseline | 81.19 (11.17)
  Diastolic blood pressure at 2 months | 79.49 (9.36)

3. Secondary Outcome: Self-report Adherence to Medication
Description: Self-report adherence to medication will be measured based on qualitative analysis of the Krousel-Wood Medication Adherence Scale 4. The subject will complete the survey twice, at baseline visit and at the end of study visit. The score range is 0 to 4 with a higher score indicating worse adherence, and a lower score indicating better adherence.
Time Frame: Baseline, 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Group
Number analyzed (Participants) | 36
units on a scale
  Adherence at baseline | 2.19 (0.86)
  Adherence at 2 months | 1.58 (0.87)

4. Secondary Outcome: Change in Systolic and Diastolic Blood Pressure Done by the Participant
Description: The subjects were asked to perform the self measured systolic and diastolic blood pressure readings at home everyday. There is increased accuracy of obtaining 7-day average systolic blood pressure (SBP) and diastolic blood pressure (DBP) measurements to assess blood pressure lowering, these measurements were obtained during the first and last week of the study. The investigators used the first and last 7-day average to calculate this outcome measure.
Time Frame: First week of the study, Last week of the study
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Patient Group
Number analyzed (Participants) | 36
mmHg
  Systolic blood pressure (first 7-day average) | 131.21 (12.34)
  Systolic blood pressure (last 7-day average) | 127.00 (11.54)
  Diastolic blood pressure (first 7-day average) | 78.07 (6.45)
  Diastolic blood pressure (last 7-day average) | 77.00 (8.77)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Patient Group
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/73/NCT05074173/Prot_SAP_000.pdf